CLINICAL TRIAL: NCT02337478
Title: An Open Label, Phase II Study of the Feasibility and Efficacy of Vincristine Sulfate Liposome Injection in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Vincristine Sulfate Liposome in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped early due to futility.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00030674; NCI-2014-02535 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 22214 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vincristine sulfate liposome) (Experimental): Patients receive vincristine sulfate liposome via injection on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Vincristine Sulfate Liposome; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Vincristine Sulfate Liposome — Given via injection
  Other Names: liposomal vincristine; Marqibo; vincristine liposomal; vincristine sulfate liposome injection
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies how well vincristine sulfate liposome works in treating patients with acute myeloid leukemia that has returned after a period of improvement or has not responded to previous treatment. Drugs used in chemotherapy, such as vincristine sulfate liposome, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Liposomal encapsulation prolongs bioavailability (proportion of drug that enters the circulation when introduced into the body) of vincristine sulfate, and may increase its delivery to cancer cells with fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of administering vincristine sulfate liposome injection (VSLI) to relapsed or refractory acute myeloid leukemia (AML) patients having failed, refused or not a candidate for at least one chemotherapy salvage regimen.

II. To observe the hematologic improvement-rate of VSLI in this patient population.

SECONDARY OBJECTIVES:

I. To observe the overall survival of patients treated with VSLI. II. To observe the response rate (complete remission [CR], complete remission with incomplete count recovery [CRi], partial response [PR], and morphologic leukemia free state [MLFS]) of VSLI in this patient population.

OUTLINE:

Patients receive vincristine sulfate liposome via injection on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented relapsed and/or refractory acute myeloid leukemia
* Patients must be ineligible for, refused or having failed at least one previous salvage regimen
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study period, unless documentation of infertility exists
* Mentally competent, ability to understand and willingness to sign the informed consent form
* No serious medical illness that would potentially increase patients' risk for toxicity
* No active central nervous system (CNS) disease
* No active uncontrolled bleeding/bleeding diathesis
* No condition or abnormality which may, in the opinion of the investigator, compromise the safety of the patient
* No unwillingness or inability to follow protocol requirements
* No evidence of ongoing, uncontrolled infection
* No requirement for immediate palliative treatment of any kind including surgery
* No option for immediate bone marrow transplant unless patient refuses this therapy
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) =< 3 x upper normal limit (UNL), alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3 x UNL
* Bilirubin =< 3 x UNL
* Glomerular filtration rate (GFR) > 50 ml/min/1.72 m^2 or creatinine < 2 g/dL

Exclusion Criteria:

* Serious medical illness or severe debilitating pulmonary disease that would potentially increase the patients' risk for toxicity
* Patients with persistent grade 3 or higher prior vincristine (VCR) (vincristine sulfate)-related neuropathy
* Patients with active central nervous system (CNS) disease
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* Pregnant women, or women of child-bearing potential not using reliable means of contraception
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Evidence of ongoing, uncontrolled infection
* Patients with known human immunodeficiency virus (HIV) infection
* Requirement for immediate palliative treatment of any kind including surgery
* Evidence of inadequate hepatic function (aspartate aminotransferase [AST/SGOT] =< 3 x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] =< 3 x UNL [=< 5 x ULN if liver metastases present], bilirubin =< 1.5 x UNL)
* Evidence of inadequate renal function (creatinine > 2 g/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pardee, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Vincristine Sulfate Liposome)
Started | 5
Completed | 0
Not Completed | 5
Not completed — Lack of Efficacy | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vincristine Sulfate Liposome)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Able to Complete Two or More Courses of Therapy Regardless of Dose Modifications
Time Frame: Up to 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vincristine Sulfate Liposome)
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Response Rate (CR, CRi, PR, and MLFS)
Description: Confidence intervals will be calculated around the estimates of the response rate (CR, CRi, PR, and MLFS) of VSLI. Assuming a response rate of 0.1, with 39 participants, 95 percent confidence intervals with a 0.09 margin of error (0.01, 0.19) or a margin of error of 0.16 around a response rate of 0.5 will be created.
  (Complete remission (CR) bone marrow blasts <5%, absence of blasts with Auer rods; absence of extramedullary disease, absolute neutrophil count >1,000, platelet count >100,000, independence of red cell transfusions; Complete remission with incomplete recovery (CRi) all complete remission except for residual neutropenia or thrombocytopenia; partial remission (PR), decrease of bone marrow blast to 5-25%, decrease of pre-treatment bone marrow blast by at least 50%; morphologic leukemia-free state (MLFS) Bone marrow blasts <5%, absence of Aeur rods, absence of extramedullary disease, no hematologic recovery required).
Time Frame: Up to 6 months after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vincristine Sulfate Liposome)
Number analyzed (Participants) | 5
Participants
  No response | 5
  Complete response | 0
  Complete reponse (incomplete) | 0
  Partial response | 0
  Morphologic leukemia free state | 0

3. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimation will be used to analyze overall survival.
Time Frame: Up to 6 months after completion of therapy
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vincristine Sulfate Liposome)
Number analyzed (Participants) | 5
months | 1.5 [1.0 to 11.6]

ADVERSE EVENTS:
Time Frame: Over 6 months
Description: Adverse events were captured for 8 days after the last dose of Vincristine Sulfate Liposome Injection (VSLI). Serious adverse events includes all Grade 5 and unexpected Grade 4 toxicities
Arm/Group | Treatment (Vincristine Sulfate Liposome)
All-Cause Mortality (participants affected / at risk) | 5/5
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vincristine Sulfate Liposome) (N=5)
Death (General disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vincristine Sulfate Liposome) (N=5)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Cardiac disorders, other (Cardiac disorders) | 2 (2)
Cardiac troponin I increased (Investigations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Chills (General disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema limbs (General disorders) | 4 (4)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorders, other (Gastrointestinal disorders) | 1 (2)
General disorders and administration site conditions - Other (General disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6)
Headache (Nervous system disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphastemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Investigations - other (Investigations) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (5)
Mucosal infection (Infections and infestations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Nervous system disorders Other (Nervous system disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 4 (5)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Platelet count decreased (Investigations) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Reproductive system and breast disorder - other (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorder - other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Scleral disorder (Eye disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 3 (3)
Skin infection (Infections and infestations) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Weight loss (Metabolism and nutrition disorders) | 3 (3)
White blood cell decreased (Investigations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes